CLINICAL TRIAL: NCT03234257
Title: Evaluation of the Carotid Plaque Stability by Ultrafast-ultrasound Imaging (UF)
Acronym: UF-Plaques
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: French Cardiology Society (Other)
Collaborators: INSERM U979 (Institut Langevin) (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2016-03
Record Dates: First submitted 2017-07-10; First posted 2017-07-31 (Actual); Last update posted 2021-08-09 (Actual); Status verified 2021-08

CONDITIONS: Carotid Stenosis
Keywords: Carotid stenosis; stiffness; ultrafast ultrasound imaging; Plaque stability
MeSH Terms: conditions — Carotid Stenosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- patients with carotid stenosis. (Other): asymptomatic patients with carotid stenosis.
  Interventions: Device: UF-ultrasound

INTERVENTIONS:
Device: UF-ultrasound — the carotid plaque stability by UF in order to improve the stroke prediction in case of asymptomatic stenosis. A UF-ultrasound approach is a non-irradiating, easily accessible, and low cost technique

SUMMARY:
Unstable plaques are characterized by lower segmental stiffness and intimal neovascularization compared to stable plaques. Our objective is to determine the capacity of the elastographic parameters obtained by the UF to discriminate the unstable to the stable plaques. We hope to improve the stroke prediction in asymptomatic patients with carotid stenosis.

DETAILED DESCRIPTION:
Context

Stroke is the second leading cause of death in the Western world and the leading cause of major disability in the long term. About 15% of strokes are secondary to thrombosis or embolization of an unstable atherosclerotic plaque of the carotid bifurcation. In these symptomatic patients, the degree of carotid stenosis is correlated with the risk of early recurrence. In patients with stenosis (NASCET)> 70%, endarterectomy is an intervention aimed at removing the carotid plaque to prevent stroke. In asymptomatic patients, the degree of stenosis is a limited predictive factor and a better risk stratification is required to assess the degree of the plaque vulnerability. The therapeutic decision towards endarterectomy in addition to drug therapy is debated because of a variable benefit/ risk balance. Several imaging parameters were studied: anfractuosity, heterogeneity, and vascularization of the plaque for example, without allowing a modification of the current recommendations. Our objective is to improve the evaluation of the risk of stroke by the fine characterization of the carotid stenosis to help the medical decision. We want to evaluate a new ultrasound imaging technology called Ultrafast ultrasound imaging (UF). Ultrasound has the advantage of being a non-irradiating, low-cost easily accessible.

Hypotheses

Unstable plaques are characterized by lower segmental stiffness and intimal neovascularization compared to stable plaques. Our objective is to determine the capacity of the elastographic parameters obtained by the UF to discriminate the unstable to the stable plaques. We hope to improve the stroke prediction in asymptomatic patients with carotid stenosis.

Innovative aspects

The originality of the approach is the use of an advanced imaging technique, UF, developed by the Langevin Institute with Mathias Fink, and already validated in the study of arterial stiffness with pulse wave analysis .

This project for the application of UF in atherosclerotic plaques stems from the ability to analyze the biomechanical properties of tissues by ultrasound elastography, already developed in the breast, liver and thyroid. Not only does UF determine the tissue stiffness expressed in kPa (Young's modulus) of the arterial wall and therefore of the carotid plaque, but UF also offers the possibility of establishing a rigidity mapping at the μm3 scale And therefore to approach the variability of the rigidity inside the plaque.

Moreover, following the recent development of the Doppler UF by the Langevin Institute, the capabilities of this tool in the precise detection of microvascular flows make it a cutting-edge tool adapted to the study of the vascularization of the carotid plaque As well as the study of the hemodynamic shear stresses that apply to the surface of the plaque.

Objective

Our objective is the development and validation of informative biomarkers of the carotid plaque stability by UF in order to improve the stroke prediction in case of asymptomatic stenosis. A UF-ultrasound approach is a non-irradiating, easily accessible, and low cost technique.

The primary objective of this study is:

- to demonstrate a significant difference in the local stiffness measurement using UF between the stable and unstable plaques, according to the histological criteria.

The secondary objectives are:

1. to compare the stiffness between plaque and its adjacent arterial segments.
2. to show a correlation between the plaque's stiffness and the histological quantification of the fibrous tissue.
3. to demonstrate a correlation between the elasticity of the plaque and the histological quantification of the calcifications.
4. compare the quantification of vascularization by UF Doppler with the number of neovessels histologically quantified
5. To compare the quantification of the wall shear stress evaluated by UF Doppler between stable and unstable plaque.
6. to compare all the different parameters used to evaluated the plaque's stability, but depending on whether or not the carotid stenosis is symptomatic.

ELIGIBILITY:
Inclusion Criteria:

* Adults over 18 years, referred to H.E.G.P for carotid endarterectomy,
* beneficiaries of a social security scheme,
* having received research information and signed the consent form.

Exclusion Criteria:

* Non-atherosclerotic carotid stenosis (post-radiation stenosis)
* No social security coverage

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2017-05-18 (Actual); Primary Completion 2019-05-05 (Actual); Study Completion 2020-09-30 (Actual)

PRIMARY OUTCOMES:
local stiffness measurement | the day of enrollment
  demonstrate a significant difference in the local stiffness measurement using UF between the stable and unstable plaques, according to the histological criteria.

SECONDARY OUTCOMES:
stiffness between plaque and its adjacent arterial segments | The day of enrollment.
  compare the stiffness between plaque and its adjacent arterial segmentsThe local arterial stiffness (for plaque and its adjacent segments) is evaluated by shear wave imaging (SWE) with the Aixplorer® (SuperSonic© Imaging). Dedicated SWE sequences provide a mapping of local stiffness. The value of the stiffness retained is the average of the region fixed by contouring the plate and the adjacent segments on the B-mode image.
correlation between the plaque's stiffness and the histological quantification of the fibrous tissue. | at the end of the study (5 months)
  show a correlation between the plaque's stiffness and the histological quantification of the fibrous tissue.
correlation between the elasticity of the plaque and the histological quantification of the calcifications | The quantification of the fibrous tissue is carried out in a semi-quantitative manner by a suitable scale, which will be filled in the histological analysis
  to demonstrate a correlation between the elasticity of the plaque and the histological quantification of the calcifications.The quantification of the fibrous tissue is carried out in a semi-quantitative manner by a suitable scale, which will be filled in the histological analysis
the quantification of vascularization by UF Doppler with the number of neovessels histologically quantified | the day of enrollment
  compare the quantification of vascularization by UF Doppler with the number of neovessels histologically quantified. The quantification of the calcifications is carried out in a semi-quantitative manner by a suitable scale, which will be filled in the histological analysis
the quantification of the wall shear stress evaluated by UF Doppler between stable and unstable plaque. | the day of enrollment
  To compare the quantification of the wall shear stress evaluated by UF Doppler between stable and unstable plaque.The quantification of wall shear stress is done using the UF Doppler mode. This is the measure of the average speed of the carotid flow, in contact with the plaque.
compare all the different parameters used to evaluated the plaque's stability, but depending on whether or not the carotid stenosis is symptomatic | the day of enrollment
  to compare all the different parameters used to evaluated the plaque's stability, but depending on whether or not the carotid stenosis is symptomatic

CONTACTS AND LOCATIONS:
Overall Officials: Emmanuel MESSAS, Principal Investigator — emmanuel.messas@aphp.fr
Locations (1):
- Hopital Europeen Georges Pompidou, Paris, France

REFERENCES:
- [Derived] Goudot G, Sitruk J, Jimenez A, Julia P, Khider L, Alsac JM, El Batti S, Bruneval P, Amemyia K, Pedreira O, Mortelette H, Calvet D, Tanter M, Mirault T, Pernot M, Messas E. Carotid Plaque Vulnerability Assessed by Combined Shear Wave Elastography and Ultrafast Doppler Compared to Histology. Transl Stroke Res. 2022 Feb;13(1):100-111. doi: 10.1007/s12975-021-00920-6. Epub 2021 Jun 28. PMID 34181190